CLINICAL TRIAL: NCT06727279
Title: Assessment of Tolerability of Specialized Foods of Vegetable Proteins and Their Influence on Lipid Profile in Patients With Non-alcoholic Fatty Liver Disease
Brief Title: Assessment of Tolerability of Specialized Food Products Made Out of Vegetable Protein and Their Influence on Lipid Profile in Patients With Non-alcoholic Fatty Liver Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology (Other)
Collaborators: Group of companies EFKO (Unknown); Russian Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: OGIG-19-76-30014/2024-2MB; 19-76-30014-P (Other Grant/Funding Number: Russian Science Foundation)
Record Dates: First submitted 2024-12-06; First posted 2024-12-10 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Non-alcoholic Fatty Liver Disease NAFLD
Keywords: non-alcoholic fatty liver disease; vegetable protein; specialized foods; plant-based meat analogs; meat substitutes; tolerability
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Chicken-flavoured plant-based meat analogs will be used in this study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- plant-based meat analog (Experimental): Patients with non-alcoholic fatty liver disease will receive iso-caloric diet with modified fat and protein content: 18.8 g/day animal proteins a day will be substituted by 13.0 g/day vegetable protein; 6.0 g/day animal fat will be substituted by 19.1 g/day vegetable fat. This modification undermines substitution of a portion of meat product made of standard (animal) meat (cutlet or schnitzel) by plant-based analog, based on soy-bean source. The taste will be masked by natural food flavoring (taste of chicken).
  Interventions: Other: Specialized food - Plant-Based Meat Analog
- Control - standard iso-calorie diet (Placebo Comparator): Iso-calorie diet (based on resting energy expenditures measurements) is provided to subjects with non-alcoholic fatty liver disease
  Interventions: Other: standard isocalorie diet

INTERVENTIONS:
Other: Specialized food - Plant-Based Meat Analog — Experimental group receives specialized food made of plant-based (soy) meat analog. A portion of standard (animal) meat in a daily ration of the enrolled subjects is substituted by plant-based analog.
  Arms: plant-based meat analog
Other: standard isocalorie diet — Isocalorie (based on resting energy expenditures measurements) diet is provided to subjects of the control group with no modification of the protein and fat content
  Arms: Control - standard iso-calorie diet

SUMMARY:
To this single-centre randomized controlled comparative study it is planned to enroll 50 patients with non-alcoholic fatty liver disease. All these subjects will receive standard isocaloric diet for 14 days. Subjects of the main group will receive vegetable protein-and-fat cutlet or schnitzel insted of the same amount of standard (animal meat based) cutlet or schnitzel. Subjects of the control group will receive standard diet, with cutlets or schnitzels made of animal meat. It is planned to make repeated measurements of serum lipid profile and assess general well-being and tolerability of newly developed product compared to regular meal

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate;
* Confirmed diagnosis of non-alcoholic fatty liver disease based on EASL guidelines.

Exclusion Criteria:

* Pregnancy and breastfeeding;
* excessive alcohol intake (>20 g/day women and >30 g/day men)
* Liver cirrhosis based on liver histology, or liver stiffness measurement (LSM > or =14 kPa by Fibroscan), or APRI > or= 1; or BARD score > or = 2.
* Chronic heart failure (I-IV class by NYHA).
* Past bariatric surgery.
* Clinically relevant acute cardiovascular event within 6 months prior to screening.
* Uncontrolled arterial hypertension despite optimal anti-hypertensive therapy.
* Diabetes mellitus type 1.
* Serum glycated hemoglobin [HbA1c] concentrations >9.0%.
* Hypersensitivity to the studied product or any of its components.
* The intake of any medications that may affect the absorption, distribution, metabolism or excretion of investigational products or may lead to the induction or inhibition of microsomal enzymes (for example, indomethacin) - from the moment of randomization to the end of treatment.
* Any medical conditions that may significantly affect life expectancy, including known cancers;
* Any clinically significant immunological, endocrine, haematological, gastrointestinal, neurological or psychiatric diseases;
* Mental instability or incapacity, which may impact the ability to give informed consent, take part in the study, or affect the ability to comply with study protocol requirements.
* Positive test for to human immunodeficiency virus antibodies .
* Aspartate aminotransferase (AST) and/or ALT >10 x upper normal limits.
* conjugated bilirubin > 26 mcmol/l (patients with Gilbert's disease are allowed to the study).
* International normalized ratio >1.40.
* Platelet count <100 x10^9/L due related to portal hypertension.
* Clinically relevant renal dysfunction, including nephrotic syndrome, chronic kidney disease (determined based on the estimated glomerular filtration rate [eGFR] less than 60 ml/min/1.73 m^2).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
cholesterol | baseline and day 14
  serum cholesterol change
Low-density lipoproteins | baseline and day 14
  Serum concentrations of low-density lipoproteins change
High-density lipoproteins | baseline and day 14
  Serum concentration of HDLP change
triglycerides | baseline and day 14
  Serum concentration of triglycerides change
C-reactive protein | baseline and day 14
  Serum concentration of C-reactive protein change
urea | baseline and day 14
  serum concentration of urea change
stool form | baseline and day 14
  Stool form change assessed with standard Bristol stool scale. Type 1 is characterized by separate hard lumps, hard to pass; this often observed in constipation; Type 4 - looks like a sausage or snake, smooth and soft (normal); Type 7 - watery, entirely liquid stool, observed in diarrhea; Mean values of stool forms by previous 7 days at baseline and on day 14 will be assessed to reflect a "change".
Organoleptic qualities of the developed products | baseline and day 14
  Organoleptic assessment with the use of visual analogue scales (taste, colour, scent, texture) is to be used.
stool frequency | baseline and day 14
  Mean stool frequency a day will be assessed at baseline and at the end of the study period to detect possible "change" in bowel habits related to product use

CONTACTS AND LOCATIONS:
Overall Officials: Vasily Isakov, MD, PhD, Professor, Study Chair — Federal Research Center of Nutrition&Biotechnology

IPD SHARING:
Plan to Share IPD: Yes
Data may be shared upon reasonable request to principal investigator
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 5 years after study completion